CLINICAL TRIAL: NCT01282866
Title: Hair Count Reduction Verification Study With the LightSheer Duet HS Handpiece
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM- ABU-LSDuet-08-001
Record Dates: First submitted 2011-01-09; First posted 2011-01-25 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2014-01

CONDITIONS: Hair Removal

ARMS (1):
- HS treatment (Experimental): Treatment with HS handpiece
  Interventions: Device: LightSheer Duet

INTERVENTIONS:
Device: LightSheer Duet — LightSheer Duet HS handpiece

SUMMARY:
The objective of this clinical study is to verify hair count reduction, associated comfort/discomfort and treatment time using the LightSheer Duet System with the High Speed (HS) handpieces for temporary hair removal and permanent hair reduction. It is anticipated that the larger treatment size of the HS handpiece will result in faster treatment of larger areas; and that the lower energy levels will result in greater comfort.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult, female, 18 years of age or older with skin type I-IV;
2. Having at least one suitable treatment area for hair removal with brown hair;
3. Able and willing to comply with the treatment/follow-up schedule and requirements;
4. Able to read, understand and provide written Informed Consent.
5. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to market preference test enrollment and throughout the course of the study treatment.

Exclusion Criteria:

1. Showing symptoms of hormonal disorders, as per the Investigator's discretion;
2. Use of oral isotretinoin (Accutane®) within 6 months
3. Prior skin treatment with laser or other devices on the same treated areas prior to study enrollment or during the course of the study;
4. History of keloid formation or poor wound healing in a previously injured skin area;
5. Significant skin conditions affecting treated area or inflammatory skin conditions;
6. Open laceration, abrasion, active cold sores or herpes sores on area to be treated;
7. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications;
8. Having a history of bleeding disorder or taking anticoagulation medications before the washout period, per the package insert, and at the physician's discretion;
9. Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the area to be treated, personal history of melanoma;
10. Significant concurrent illness, such as diabetes, lupus, epilepsy or cardiac disorders, which might be aggravated as a result of treatment;
11. Unable or unlikely to refrain from tanning, including the use of tanning booths, tanning spray or cream, during the course of the evaluation;
12. Tattoos in the treatment areas;
13. Dysplastic nevi in the treatment areas;
14. Participation in a study of another device or drug within 3 month prior to study enrollment or during this study, and as per the Investigator's careful discretion, as long as not contradictory to any of the above criteria;
15. Mentally incompetent, prisoner or evidence of active substance or alcohol abuse;
16. Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or for the study personnel) to treat the subject as part of this research study;
17. Allergy or history of an allergy to any topical anesthetic used;
18. Pregnant, expectation of pregnancy, postpartum (<3 months) or nursing (<6 weeks);
19. History of livedo reticularis, an autoimmune vascular disease;
20. Hypersensitivity at the treatment site to any agents, solutions, or gel used in the treatment (applies to ET handpiece only), if no alternative exists;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Laser & Skin Surgery Medical Group Inc, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- HS Treatment: Treatment with the LightSheer Duet laser HS handpiece:
  Treatment parameters: Fluence: 9-12J/cm^2, pulse duration: 30 to 70ms,medium to low vacuum levels.
  All patients were treated in the Axilla area.
Period: Overall Study
Arm/Group | HS Treatment
Started | 35
Completed | 34
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: The power calculation proposed a sample of 35 participants to be sufficient to obtain qualitative assessment of hair removal, as well as the qualitative assessment of treatment time and pain experienced during treatment with the LightSheer Duet HS handpiece.
Arm/Group | HS Treatment
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Hair Count
Description: The hair at the treatment area is counted at Baseline and 6 months following the last treatment.
  Hair clearance is determined by the percentage of Hair left 6 months following the last treatment compared to the hair number at baseline.
Time Frame: 6 month following last treatment
Measure: Mean (Standard Deviation); unit: percentage of hair clearance
Groups:
- HS Treatment: Treatment with the LightSheer Duet laser HS handpiece:
  Treatment parameters: Fluence: 9-12J/cm2, pulse duration: 30 to 70ms,medium to low vacuum levels.
  All patients were treated in the Axilla area.
Arm/Group | HS Treatment
Number analyzed (Participants) | 34
percentage of hair clearance | 54 (24)
Statistical Analysis 1: Comparison: HS Treatment; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Treatment Time
Description: The treatment time was measured for each participant on each and every visit. The result is presented as mean of all treatment time from all of the visits and all of the participants.
Time Frame: Each treatment
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | HS Treatment
Number analyzed (Participants) | 34
minutes | 3.5 (2.7)

3. Secondary Outcome: Level of Comfort Associated With Treatment
Time Frame: Each treatment
Reporting Status: Not Posted

4. Secondary Outcome: Hair Count
Description: The hair at the treatment area is counted at Baseline and 15 months following the last treatment.
  Hair clearance is determined by the percentage of Hair left 15 months following the last treatment compared to the hair number at baseline.
Time Frame: 15 month following last treatment
Population: The number of participants who completed 15 months follow up was 23 out of 35.
Measure: Mean (Standard Deviation); unit: percentage of hair clearance
Arm/Group | HS Treatment
Number analyzed (Participants) | 23
percentage of hair clearance | 42 (25)

ADVERSE EVENTS:
Arm/Group | HS Treatment
Serious Adverse Events (participants affected / at risk) | 1/35
Other Adverse Events (participants affected / at risk) | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HS Treatment (N=35)
injured ankle (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No